CLINICAL TRIAL: NCT05563194
Title: Exploring the Potential of 'JIA Toolbox' in Improving the Independence and Functional Ability of Children and Young People (CYP) With Juvenile Idiopathic Arthritis (JIA)
Brief Title: Proof-of-concept Study of 'JIA Toolbox' for Children and Young People (CYP) With Juvenile Idiopathic Arthritis (JIA)
Acronym: JIA Toolbox
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SCH-2628
Record Dates: First submitted 2022-09-21; First posted 2022-10-03 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Rheumatologic Disease
MeSH Terms: conditions — Collagen Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Children and young people with a diagnosis of Juvenile Idiopathic arthritis (Experimental): Single arm study where all participants will receive the three prototype interventions.
  Interventions: Device: Heating prototype (Prototype 1); Device: Physio tool (Prototype 2); Device: Communication tool (Prototype 3)

INTERVENTIONS:
Device: Heating prototype (Prototype 1) — A wearable that heats and vibrates to help distract from pain. It can be wrapped around any joint with temperature and vibration settings allowing CYP to set the device to their needs.
Device: Physio tool (Prototype 2) — A motivational physiotherapy tool that incrementally lights up as the CYP do their prescribed stretches, emphasising a sense of progression and making it a more engaging activity.
Device: Communication tool (Prototype 3) — A wearable to help communication in the classroom between the teacher and pupil. The child can alert the teacher if they need help, through vibration, without attracting the attention of their classmates, reducing embarrassment.

SUMMARY:
This project aims to further develop and conduct a 'real-world' proof-of-concept assessment of a suite of three products, known as the 'JIA Toolbox', that collectively aim to improve CYP's independence and functional ability

'JIA Toolbox' targets key unmet needs identified by stakeholders during our previous work. Each prototype (Appendix1) addresses a specific unmet need:

1. Prototype-1: Pain which stops CYP doing the things they love;
2. Prototype-2: Difficulty for healthcare professionals (HCPs) to motivate CYP to do stretches;
3. Prototype-3: Communication difficulties between teachers and CYP

The project is at a stage where the prototypes need their potential value assessed through a proof-of-concept study. A co-design approach, involving CYP with JIA, their parents, their teachers and HCPs, will be maintained throughout to ensure the outcomes are meaningful. This study will begin with co-design workshops to develop the current prototypes further, followed by a qualitative study assessing the real-world usability, acceptability and potential impacts of these prototypes; testing them with real users in their homes. The project aims to make a positive contribution to CYP with JIA by improving their independence and functional ability through co-designed therapeutic interventions.

DETAILED DESCRIPTION:
Juvenile Idiopathic Arthritis (JIA) is a long-term rheumatic disease affecting approximately 15,000 children and young people (CYP) in the UK [1] with 1,000-1,500 new diagnoses/year. JIA causes ongoing/long-term joint inflammation, pain, and stiffness, making everyday activities difficult. JIA has been shown to impact physical, social, emotional, and educational development. Products exist to aid tasks such as writing, washing, and eating. However, a survey we conducted in 2018 showed that CYP with JIA find these products difficult to use, stigmatising, and patronising. Furthermore, these products often neglect to consider the wider stakeholder network and how their support, or lack of it, impacts the child's overall wellbeing.

This project aims to further develop and conduct a 'real-world' proof-of-concept assessment of a suite of three products, known as the 'JIA Toolbox', that collectively aim to improve CYP's independence and functional ability

'JIA Toolbox' targets key unmet needs identified by stakeholders during our previous work. Each prototype (Appendix1) addresses a specific unmet need:

1. Prototype-1: Pain which stops CYP doing the things they love;
2. Prototype-2: Difficulty for healthcare professionals (HCPs) to motivate CYP to do stretches;
3. Prototype-3: Communication difficulties between teachers and CYP

The project is at a stage where the prototypes need their potential value assessed through a proof-of-concept study. A co-design approach, involving CYP with JIA, their parents, their teachers and HCPs, will be maintained throughout to ensure the outcomes are meaningful. This study will begin with co-design workshops to develop the current prototypes further, followed by a qualitative study assessing the real-world usability, acceptability and potential impacts of these prototypes; testing them with real users in their homes. The project aims to make a positive contribution to CYP with JIA by improving their independence and functional ability through co-designed therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* Aged 7- 16 years (minimum age is 7 to ensure participants can adequately engage with the prototypes and describe their experience)
* Diagnosis of JIA
* Currently managed within SCH Rheumatology Service
* Fluent in verbal and written English
* Access to a computer with an internet connection to facilitate virtual co-design workshops due to the COVID-19 pandemic

Exclusion Criteria:

* Aged <7 years or >16 years
* Non-fluent in verbal and written English
* Diagnosis of autistic spectrum disorder (ASD)
* Children with medically unexplained pain, pain amplification syndromes or other pain disorder
* Co-existing joint or muscle disorder other than JIA

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Change in self-management of JIA | Baseline, Week 9
  Changes in the participants ability to self-manage their condition independently and confidently. Assessed through daily questionnaires throughout the duration of the study, data (frequency of use, settings chosen) from the prototypes, and a post-intervention interview with participants.
Change in functional ability | Baseline, Week 9
  Changes in ability across physical, emotional, social and educational spheres. Assessed through daily questionnaires throughout the duration of the study, data (frequency of use, settings chosen) from the prototypes, and a post-intervention interview with participants.
Change in physio adherence | Baseline, Week 9
  Change in frequency of participants undertaking recommended physio stretches. Assessed through daily questionnaires throughout the duration of the study, data (frequency of use, settings chosen) from the prototypes, and a post-intervention interview with participants
Change in pain-management | Baseline, Week 9
  Change in participants ability to manage joint pain during a flare up using prototype 1. Assessed through daily questionnaires throughout the duration of the study, data on prototype 1 (frequency of use, settings chosen), and a post-intervention interview with participants.

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Ankeny, Study Director — Sheffiled Hallam University
Locations (1):
- Sheffield Children's NHS Foundation Trust, Sheffield, United Kingdom